CLINICAL TRIAL: NCT06507956
Title: Physical Activity Profile and Sedentary Behaviour in Adults With Cystic Fibrosis
Acronym: ACTIVMUCO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1132; 2024-A01077-40 (Other: ID-RCB)
Record Dates: First submitted 2024-07-10; First posted 2024-07-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Exercise; Sedentary lifestyle
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with cystic fibrosis followed at Hôpital Lyon Sud's cystic fibrosis center-single-arm study.
  Interventions: Other: Characterize the physical activity and sedentary lifestyle profile of adults with cystic fibrosis

INTERVENTIONS:
Other: Characterize the physical activity and sedentary lifestyle profile of adults with cystic fibrosis — Eligible patients will be presented with the study during a routine care visit CF center, at the end of a physiotherapy, adapted physical activity or nurse session, in accordance with the schedule for the day's visit, with no changes induced by this study. After sufficient time for reflection, patients agreeing to participate will be given self-questionnaires. From this visit, a proposal to participate at V2 will be made only to the inactive and/or hight sedentary patients on the ONAPS-PAQ questionnaire, under elexacaftor-tezacaftor-ivacaftor (ETI). Volunteers will know their participation in either actimetry or a qualitative interview following a draw. At V2, 40 patients will be offered a 7-day longitudinal follow-up by actimetry, and between 10 to 15 patients will take part in an qualitative semi-structured interview identifying motivational barriers and levers for action. At V3, patients monitored by actimetry will be invited to return their actimeter by postage-paid mail.

SUMMARY:
Cystic fibrosis is a multisystem genetic disease whose severity, linked to the nature of the mutation in the gene carried, is linked to respiratory impairment, which determines the vital prognosis.

Considerable progress has been made in the management of this disease, amplified in recent years by the arrival of CFTR (cystic fibrosis transmembrane conductance regulator) modulator drugs, and in particular the triple treatment combination of elexacaftor-tezacaftor-ivacaftor (ETI). This modulator therapy improves clinical condition, particularly respiratory, and transforms quality of life and prognosis for some patients. Faced with this clinical improvement, practices and care paths are adapting. Professionals will have to cope with the emergence of new clinical conditions linked to the ageing of this at-risk population and the functional decline due to a sedentary lifestyle and age.

The working hypothesis is that a better understanding of the physical activity and sedentary lifestyle profiles of the adult population with cystic fibrosis, and in particular the characterization of the profile of inactive and high sedentary patients under ETI, will enable us to identify and target patients whose lifestyle habits reflect a greater health risk, and for whom care by rehabilitators and adapted physical activity (APA) teachers and personalized advice could be put in place.

The aim of this study is to characterize the physical activity and sedentary profile of adults with cystic fibrosis.

ACTIVMUCO is an observational, cross-sectional, single-center study. A subgroup of adults with high sedentary and inactive under ETI will be studied more specifically by actimetry (prospective follow-up) and interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) of legal age,
* Patients with cystic fibrosis (CF) regularly followed at Hôpital Lyon Sud's cystic fibrosis center, who volunteered to take part in the study.

Exclusion Criteria:

* People who, due to the presence of co-morbidities, do not have motor and cognitive skills compatible with independent walking or orthostatic physical activity.
* People whose clinical situation contraindicates the practice of adapted physical activity
* Pregnant women
* People who do not have the intellectual or linguistic capacity to understand the questionnaires
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults under legal protection (guardianship, curatorship).
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants (male or female of legal age, with cystic fibrosis - CF) are recruited from the active file of adult patients followed at the CF Reference Center of Hôpital Lyon Sud, from the Rhône-Alpes region of France. They must be volunteers to participate in the study. The study ACTIVMUCO is carried out at the time of the patient's scheduled visit, on site, without impacting the dynamics of the care pathway, on an active file of around 430 patients. The regularity of these outpatient visits to the CF center is between 1 and 4 times a year, depending on the patient's clinical condition. The number of patients to be recruited is 270. The number of patients followed regularly over the past year was 434, including 85 transplant patients and 20 new patients. Over the 12-month recruitment period, the department estimates that around 80% of patients followed will actually come for day hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity and sedentary levels will be quantified by the weekly time calculation of moderate physical activity | For each subject : day 1 for the cross-sectional questionnaire study - 3 months to 6 months (next consultation at the CF center) and 1 week for the subgroup monitored by accelerometry
  Moderate physical activity self-reported and reported in METs (Metabolic Equivalent of Task).minutes/week on the ONAPS-PAQ questionnaire, then categorized into 3 physical activity profiles:
  1. Inactive individual
  2. Active individual
  3. Very active individual
Physical activity and sedentary levels will be quantified by the weekly time calculation of high-intensity physical activity | For each subject : day 1 for the cross-sectional questionnaire study - 3 months to 6 months (next consultation at the CF center) and 1 week for the subgroup monitored by accelerometry
  High-intensity physical activity self-reported and reported in METs (Metabolic Equivalent of Task).minutes/week on the ONAPS-PAQ questionnaire, then categorized into 3 physical activity profiles:
  1. Inactive individual
  2. Active individual
  3. Very active individual
Physical activity and sedentary levels will be quantified by the weekly time calculation of 2. Sedentary activity | For each subject : day 1 for the cross-sectional questionnaire study - 3 months to 6 months (next consultation at the CF center) and 1 week for the subgroup monitored by accelerometry
  Sedentary activity self-reported and reported in daily average (hours/day) on the ONAPS-PAQ questionnaire, then categorized into sedentary levels:
  1. Low
  2. Moderate
  3. High

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No